CLINICAL TRIAL: NCT07159451
Title: A Short-term Preoperative, Window-of-opportunity Study, Evaluating Activity and Safety of Elacestrant Monotherapy as Compared to Elacestrant + Ovarian Function Suppression (LHRH Agonist) in Premenopausal Patients With Stage I-II ER+/HER2- Breast Cancer
Brief Title: A Short-term Preoperative, Evaluating Activity and Safety of Elacestrant Monotherapy as Compared to Elacestrant + Ovarian Function Suppression (LHRH Agonist) in Premenopausal Patients With Stage I-II ER+/HER2- Breast Cancer
Acronym: POP-ELA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-520051-24-00; 2025/4053 (Other: CSET number)
Record Dates: First submitted 2025-08-19; First posted 2025-09-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: early-stage; HR+ breast cancer; breast cancer; premenopausal patients; stage I-II; ER+/HER2- breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): Patients will receive elacestrant 345 mg/daily administered orally for 4 weeks.
  Interventions: Drug: Elacestrant
- Experimental group B (Experimental): Patients will receive elacestrant 345 mg/daily administered orally for 4 weeks with leuprorelin LP 3.75 mg intramuscular Day 1 and Day 29.
  Interventions: Drug: Elacestrant; Drug: Leuprorelin

INTERVENTIONS:
Drug: Elacestrant — Patients will receive elacestrant 345 mg/daily administered orally for 4 weeks.
Drug: Leuprorelin — Patients randomized in arm B will recieve Leuprorelin at Day 1 and Day 29
  Arms: Experimental group B

SUMMARY:
A prospective randomized trial designed to evaluate the mean decrease in Ki67 after 4 weeks of elacestrant monotherapy and in combination with leuprorelin in patients with early-stage HR+ BC. This preoperative study will enroll consecutive patients with early stage HR+ BC who are not candidates for neoadjuvant chemotherapy but are eligible for short-term preoperative treatment with elacestrant, with or without leuprorelin, followed by breast surgery. A total of three dedicated Formalin-fixed paraffin embedded (FFPE) samples (mandatory for all patients), along with two frozen biopsy (only for participants at Gustave Roussy), are planned to be collected at the time of inclusion from the biopsy sample and from the surgical specimen. Blood samples will also be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be randomized in the study:

1. Aged 18 or more.
2. Signed Informed Consent Form prior to any study-specific procedure. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Patients must be affiliated to a Social Security System (or equivalent).
4. Premenopausal women ensured by checking if the women were still having regular periods over the last 6 months without any hormonal treatment or hormonal contraception or if they were irregular, FSH and estradiol levels must fall within the premenopausal range according to local laboratory definition.
5. Histologically confirmed invasive breast carcinoma, confirmed by the local pathologist, ER-positive tumor cells ≥ 10% ER staining BC and HER2- according to ASCO criteria in immunohistochemistry (IHC) and/or genomic analysis (HER2 negativity is defined as IHC 0-1+, or [IHC 2+ and in situ hybridization non-amplified]), Ki67 index by local analysis of ≥ 10% and ≤ 30% on untreated tumor tissue.
6. Clinical stage I or II according to the eight edition of the American Joint Committee on Cancer, eligible for primary breast surgery.

   Note: Multifocal and multicentric tumors are permitted if they are considered clinical stage I or II according to Eight Edition of the AJCC. Biopsy of all lesions is not necessary and is left at the description of the investigator, but endocrine therapy response must be evaluated on the same tumor
7. Available pre-treatment tru-cut biopsy evaluable.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 14 days prior to the date of randomization.
9. Women of childbearing potential have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
10. Demonstrate adequate organ function within 7 days of inclusion :

    1. Absolute neutrophil count ≥ 1.0 x 109/L
    2. Platelet count ≥ 75 x 109/L
    3. Hemoglobin ≥ 9.0 g/dL
    4. Estimated glomerular filtration rate ≥30 mL/min/1.73 m² or creatinine clearance calculated by Cockcroft-Gault equation ≥ 30 mL/min Creatinine clearance ≥ 30 mL/min for subject with creatinine levels > 1.5 x institutional upper limit of normal (ULN).
    5. Alanine aminotransferase (ALT) ≤ 2.5x upper limit of normal (ULN).
    6. Aspartate aminotransferase (AST) ≤ 3x ULN.
    7. Total bilirubin ≤ ULN or total bilirubin ≤ 1.5x ULN with direct bilirubin ≤ ULN of the laboratory in subjects with documented Gilbert's Syndrome.
    8. Potassium, sodium, calcium (corrected for albumin), magnesium, and phosphorus CTCAE v5.0 Grade ≤ 1. If Screening assessments are abnormal, chemistry assessments may be repeated up to 2 times; subjects may receive appropriate supplementation or treatment (eg, for hypercalcemia) prior to re-assessment.
    9. International normalized ratio (INR) ≤ 1.5; subjects who are receiving anticoagulation treatment which is monitored by international normalized ratio (INR) (eg, warfarin) may be allowed to participate if they have a stable INR (ie, within therapeutic range) for at least 28 days prior to the first dose of study drug, in the absence of any exclusionary medical conditions, and provided that elacestrant would be appropriate therapy for the subject.
11. Women of childbearing potential must agree to use protocol-specified method(s) of contraception during trial treatments and for at least 120 days after the last dose of trial treatments. Highly effective contraception methods include:

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Placement of a non-hormonal intrauterine device.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will not be eligible for this study.

1. Patients non-candidate for upfront breast surgery or candidate for neoadjuvant chemotherapy.
2. Any systemic therapy (e.g, chemotherapy, targeted therapy, immune-therapy) or radiotherapy for current BC before study entry.
3. Prior treatment with LHRH-agonists over the last 6 months prior to the ICF signature.
4. Any active treatment for any cancer disease.
5. Any of the following within 6 months before enrollment:

   1. Myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE v5.0 Grade ≥2,
   2. Prolonged QTcF ≥ Grade 2 (ie, > 480 msec), uncontrolled atrial fibrillation of any grade, coronary/peripheral artery bypass graft, heart failure ≥ Class II as defined by the New York Heart Association guidelines,
   3. Cerebrovascular accident including transient ischemic attack
   4. Child-Pugh Score greater than Class A,
   5. Has a known hypersensitivity (≥ Grade 3) to the components of the study therapy or its analogs.
   6. Coagulopathy or any history of coagulopathy within the past 6 months, including history of deep vein thrombosis or pulmonary embolism. However, subjects with the following conditions will be allowed to participate:
   7. Adequately treated catheter-related venous thrombosis occurring > 28 days prior to the first dose of study drug
6. Treatment with an anticoagulant, eg, warfarin or heparin, for a thrombotic event occurring > 6 months before enrollmentenrolment, or for an otherwise stable and allowed medical condition (eg, well controlled atrial fibrillation), provided dose and coagulation parameters (as defined by local standard of care) are stable for at least 28 days prior to the first dose of study drug and provided that an AI would be an appropriate therapy for the subject.
7. Known difficulty in tolerating oral medications or conditions which would impair absorption of oral medications such as: uncontrolled nausea or vomiting (ie, CTCAE ≥ Grade 3 despite antiemetic therapy), ongoing gastrointestinal obstruction/motility disorder, malabsorption syndrome, or prior gastric bypass.
8. Unable or unwilling to avoid prescription medications, over-the-counter medications, dietary/herbal supplements (eg, St. John's wort), and/or foods (eg, grapefruit, pomelos, star fruit, Seville oranges and their juices) that are moderate/strong inhibitors or inducers of CYP3A4 activity. Participation will be allowed if the medication, supplements, and/or foods are discontinued for at least 5 half-lives or 14 days (whichever is longer) prior to study entry and for the duration of the study.
9. Pregnancy or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes.
10. Any concurrent severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with compliance with study procedures or the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
11. Person deprived of their liberty or under protective custody or guardianship.
12. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
13. Patients unwilling to or unable (as assessed by the investigator) to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
To determine if 4 weeks of elacestrant monotherapy determines a non-inferior anti-proliferative effect, measured by Ki67, in comparison to elacestrant with leuprorelin in premenopausal patients with ER-positive/HER2- operable invasive BC. | Surgery

SECONDARY OUTCOMES:
Complete cell cycle arrest (CCCA) measured by Ki67 <2.7% | Surgery
Objective Response Rate | From baseline to day 29
  partial and complete response obtained as measured by MRI
Rate of pathological of partial and complete response | at surgery
Levels of estradiol | at baseline, Day 14, and Day 28 then postoperatively at 1 month
Levels of follicle-stimulating hormone (FSH) | at baseline, Day 14, and Day 28 then postoperatively at 1 month
Levels of luteinizing hormone (LH) | at baseline, Day 14, and Day 28 then postoperatively at 1 month
Incidence of treatment-emergent AEs | From enrollment until 28 days post surgery
  assessed by the national cancer institute (NCI) Common Terminology for Classification of Adverse Events (CTCAE) version 5.0,
Duration of treatment-emergent AEs | From enrollment until 28 days post surgery
  assessed by the national cancer institute (NCI) Common Terminology for Classification of Adverse Events (CTCAE) version 5.0,
Severity of treatment-emergent | From enrollment until 28 days post surgery
  AEs assessed by the national cancer institute (NCI) Common Terminology for Classification of Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No